CLINICAL TRIAL: NCT00631241
Title: Histopathologic Analysis of Parametrial Lymph Nodes as Sentinel Nodes in Patients With Cervical Cancer Undergoing Radical Hysterectomy or Radical Trachelectomy and Pelvic Lymph Node Dissection: A Feasibility Study
Brief Title: Analysis of Parametrial Lymph Nodes as Sentinel Nodes in Patients With Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0153
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Parametrial Lymph Nodes; Sentinel Nodes; Intraoperative Lymphatic Mapping; Single Photon Emission Computed Tomography; SPECT/CT
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraoperative Lymphatic Mapping (Experimental): Single Photon Emission Computed Tomography - First 3 Patients = Performed 30-45 minutes, 2-3 hours, and 20-24 hours after injections of the radioactive material or just before surgery; Remaining 17 Patients = Performed only one at a time as was found to be best based on the scans from first 3 patients. Isosulfan Blue and India ink will be injected into the cervix to help the surgeon identify the sentinel nodes by their blue color and their level of radioactivity.
  Interventions: Procedure: Single Photon Emission Computed Tomography; Procedure: Intraoperative Lymphatic Mapping

INTERVENTIONS:
Procedure: Single Photon Emission Computed Tomography — First 3 Patients = Performed 30-45 minutes, 2-3 hours, and 20-24 hours after injections of the radioactive material or just before surgery; Remaining 17 Patients = Performed only one at a time as was found to be best based on the scans from first 3 patients.
  Other Names: SPECT/CT
Procedure: Intraoperative Lymphatic Mapping — Isosulfan Blue and India ink will be injected into the cervix to help the surgeon identify the sentinel nodes by their blue color and their level of radioactivity.

SUMMARY:
The goal of this clinical research study is to find out if the parametrial nodes are "sentinel" nodes (the lymph nodes believed to be the greatest risk for the spread of cancer) and if intraoperative lymphatic mapping can identify "sentinel" lymph nodes in the parametrium (the tissue that is on either side of the cervix). Identifying these lymph nodes may help to predict the status of the remaining lymph nodes in the pelvis. This research will also determine if India Ink is safe to use with the blue dye and radioactive tracer and if it improves the process of identifying the sentinel nodes.

DETAILED DESCRIPTION:
Lymph nodes are glands that play an important part in your body's defense against infection. They are also the most common site of cancer spread in patients with cervical cancer. Intraoperative lymphatic mapping is a procedure that has been used in patients with other types of cancer to identify the "sentinel" lymph node. Researchers know that if the sentinel node does not contain cancer, then the remaining lymph nodes are almost always cancer-free.

Researchers believe that the parametrial lymph nodes (1 group of lymph nodes located in the parametrium) are the sentinel lymph nodes in patients with cervical cancer. Surgical removal of the parametrial lymph nodes is currently the only known way to accurately find out whether or not these lymph nodes have cancer in them.

Stage IA2 or IB1 cervix cancer is treated by a radical hysterectomy (removal of the uterus, cervix, and the parametrium) or radical trachelectomy (removal of the cervix and the parametrium). Pelvic lymph nodes and possibly para-aortic lymph nodes (near the aorta in the abdomen) are also removed. This procedure is called a pelvic and para-aortic lymphadenectomy.

If you agree to take part in this study, you will undergo a procedure called intraoperative lymphatic mapping. This procedure is done in the operating room. When you are asleep (under anesthesia), the surgeon will inject the cervix with a very small amount (less than one tenth of a teaspoon) of a radioactive material in 4 different places around the edge of the tumor in the cervix. This injection is given over 1-2 minutes. The cervix is then injected with 2 different blue dyes called Isosulfan Blue and India ink (about 1 1/2 teaspoons). These injections take less than 5 minutes. The surgeon will then use a special hand-held instrument for measuring radioactivity to help find the sentinel lymph nodes before and after the operation begins. During the operation, the surgeon will also visually inspect the lymph nodes to see if they are blue (stained by the blue dye and India Ink). These 2 techniques (the radioactive material and the dye and ink) will help the surgeon identify the sentinel nodes by their blue color and their level of radioactivity.

During your hospitalization or at your first clinic visit, your doctor will tell you whether or not cancer was found in the lymph nodes that were removed during surgery.

You will be taken off study if intolerable side effects occur. You will be considered off study after your first doctor's visit after the surgery.

This is an investigational study. Up to 20 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are dispositioned to undergo radical hysterectomy or radical trachelectomy and pelvic lymphadenectomy.
2. No evidence of metastases on computed tomography, magnetic resonance imaging, or PET/CT scan.
3. Patients must be good surgical candidates.
4. Patients who have signed an approved informed consent and authorization permitting release of personal health information.
5. For patients of child-bearing age, a negative serum pregnancy test within 72 hours prior to injection of radiocolloid. Child-bearing potential is defined as not post-menopausal for 12 months or no previous surgical sterilization.

Exclusion Criteria:

1. Patients with known allergies to triphenylmethane compounds or India ink.
2. Patients with a history of retroperitoneal surgery.
3. Patients with a history of pelvic irradiation.
4. Patients who had a cold knife or LEEP cone biopsy within 4 weeks of enrollment.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of Patients with sentinel lymph nodes in the parametrium | Determination during surgery (with intraoperative lymphatic mapping)
  Sentinel nodes classified according to modification of American Joint Committee on Cancer (AJCC) staging for axillary nodes from breast cancer as follows: 1) metastases present - tumor > 2.0 mm in diameter; 2) micrometastases present - tumor cell aggregates between 0.2 and 2.0 mm in diameter; 3) isolated tumor cells - individual tumor cells or aggregates <0.2 mm in diameter, usually detected by immunohistochemistry; or 4) tumor absent - no tumor cells identified in H&E (or immunohistochemically) stained sections.
  Parametrium separated from cervix/uterus by pathology then away from primary cervical lesion will be re-examined for sentinel nodes both visually & with handheld gamma counter; & all parametrial tissue will be submitted for pathologic sectioning to detect carbon particles in parametrial sentinel nodes not detected by gamma counter or direct visualization.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Frumovitz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org